CLINICAL TRIAL: NCT01144338
Title: Exenatide Study of Cardiovascular Event Lowering Trial (EXSCEL). A Randomized, Placebo Controlled Clinical Trial to Evaluate Cardiovascular Outcomes After Treatment With Exenatide Once Weekly in Patients With Type 2 Diabetes Mellitus.
Brief Title: Exenatide Study of Cardiovascular Event Lowering Trial (EXSCEL): A Trial To Evaluate Cardiovascular Outcomes After Treatment With Exenatide Once Weekly In Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5551C00003; MB001-002 (Other: Bristol Myers Squibb); BCB109 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2010-06-10; First posted 2010-06-15 (Estimated); Results first posted 2018-08-08 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide once weekly; cardiovascular; Bydureon; Amylin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exenatide Once Weekly (Experimental)
  Interventions: Drug: Exenatide Once Weekly
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide Once Weekly — Subcutaneous injection, 2 mg, administered once weekly.
  Arms: Exenatide Once Weekly
Drug: Placebo — Subcutaneous injection, matching volume of placebo, administered once weekly.
  Arms: Placebo

SUMMARY:
This study will compare the impact of including exenatide once weekly in addition to usual care vs. usual care without exenatide on major cardiovascular outcomes as measured by the primary composite endpoint of cardiovascular-related death, nonfatal myocardial infarction (MI), or nonfatal stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patient has type 2 diabetes mellitus
* Patient has an HbA1c of ≥ 6.5 % and ≤ 10.0% and is currently using one of the following treatment regimens: A) Treatment with 0-3 oral antihyperglycemic agents B) Insulin therapy, either alone or in combination with up to two oral agents
* Female patients must not be breast feeding and agree to use an effective method of contraception or must not otherwise be at risk of becoming pregnant.

Exclusion Criteria:

* Patient has a diagnosis of type 1 diabetes mellitus, or a history of ketoacidosis.
* Patient has ever been treated with an approved or investigational GLP-1 receptor agonist.
* Patient is enrolled in another experimental protocol which involves the use of an investigational drug or device, or an intervention that would interfere with the conduct of the trial.
* Patient has a planned or anticipated revascularization procedure.
* Pregnancy or planned pregnancy during the trial period.
* Patient has end-stage renal disease or an estimated glomerular filtration rate (eGFR) of <30 mL/min/1.73m2.
* Patient has a history of gastroparesis or pancreatitis.
* Personal or family history of medullary thyroid cancer or MEN2 (Multiple EndocrineNeoplasia Type 2) or calcitonin level of >40 ng/L at baseline.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14752 (Actual)
Dates: Start 2010-06-18 (Actual); Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Gustavson, PhD, Study Director — AstraZeneca; Group Director Global Clinical Research, Study Director — Bristol-Myers Squibb
Locations (507):
- United States (127):
  - Research Site, Birmingham, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Jonesboro, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Chula Vista, California
  - Research Site, Concord, California
  - Research Site, Escondido, California
  - Research Site, Fullerton, California
  - Research Site, Greenbrae, California
  - Research Site, La Mesa, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Oceanside, California
  - Research Site, Orange, California
  - Research Site, Redondo Beach, California
  - Research Site, San Diego, California
  - Research Site, Sylmar, California
  - Research Site, Torrance, California
  - Research Site, Tustin, California
  - Research Site, Victorville, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Thomaston, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Cape Coral, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Roswell, Georgia
  - Research Site, Pocatello, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Hines, Illinois
  - Research Site, Rock Island, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Gary, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Covington, Kentucky
  - Research Site, Evansville, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Auburn, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Randallstown, Maryland
  - Research Site, Rockville, Maryland
  - Research Site, Alpena, Michigan
  - Research Site, Ann Arbor, Michigan
  - Research Site, Bloomfield Hills, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Bridgeton, Missouri
  - Research Site, Chesterfield, Missouri
  - Research Site, Billings, Montana
  - Research Site, Butte, Montana
  - Research Site, Omaha, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Reno, Nevada
  - Research Site, Hamilton, New Jersey
  - Research Site, Lyons, New Jersey
  - Research Site, Margate City, New Jersey
  - Research Site, South Plainfield, New Jersey
  - Research Site, Albany, New York
  - Research Site, Manhasset, New York
  - Research Site, New York, New York
  - Research Site, North Massapequa, New York
  - Research Site, Rosedale, New York
  - Research Site, Smithtown, New York
  - Research Site, The Bronx, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Mooresville, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Salisbury, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Barberton, Ohio
  - Research Site, Canal Fulton, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Mentor, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Feasterville, Pennsylvania
  - Research Site, Lansdale, Pennsylvania
  - Research Site, Newport, Pennsylvania
  - Research Site, Penndel, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Tipton, Pennsylvania
  - Research Site, Pawtucket, Rhode Island
  - Research Site, Charleston, South Carolina
  - Research Site, Mt. Pleasant, South Carolina
  - Research Site, Murrells Inlet, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Bristol, Tennessee
  - Research Site, Chattanooga, Tennessee
  - Research Site, Jackson, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Kingsport, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, McKenzie, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Friendswood, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Webster, Texas
  - Research Site, Layton, Utah
- Argentina (12):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Capital Federal
  - Research Site, CiudadAutonoma de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Godoy Cruz
  - Research Site, Mar Del Plata Buenos Aires
  - Research Site, Rosario
  - Research Site, Salta
  - Research Site, San Miguel de Tucumán
  - Research Site, San Salvador de Jujuy
  - Research Site, Santa Rosa
- Australia (13):
  - Research Site, Adelaide
  - Research Site, Camperdown
  - Research Site, Clayton
  - Research Site, East Gosford
  - Research Site, Elizabeth Vale
  - Research Site, Fitzroy
  - Research Site, Garran
  - Research Site, Geelong
  - Research Site, Heidelberg West
  - Research Site, Meadobank
  - Research Site, Milton
  - Research Site, Parkville
  - Research Site, Sydney
- Austria (6):
  - Research Site, Feldkirch
  - Research Site, Graz
  - Research Site, Innsbruck
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Zams
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Merksem
  - Research Site, Ronse
- Brazil (11):
  - Research Site, Aparecida de Goiânia
  - Research Site, Belém
  - Research Site, Brasília
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Goiânia
  - Research Site, Marília
  - Research Site, Passo Fundo
  - Research Site, Recife
  - Research Site, São Paulo
- Bulgaria (8):
  - Research Site, Blagoevgrad
  - Research Site, Gabrovo
  - Research Site, Golenci
  - Research Site, Plovdiv
  - Research Site, Sevlievo
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Canada (23):
  - Research Site, Calgary, Alberta
  - Research Site, Delta, British Columbia
  - Research Site, New Westminster, British Columbia
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, Bridgewater, Nova Scotia
  - Research Site, Liverpool, Nova Scotia
  - Research Site, Cambridge, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kitchener, Ontario
  - Research Site, London, Ontario
  - Research Site, North York, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Smiths Falls, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Sainte-Foy, Quebec
  - Research Site, Terrebonne, Quebec
- Chile (5):
  - Research Site, Osorno
  - Research Site, Puerto Varas
  - Research Site, Santiago
  - Research Site, Temuco
  - Research Site, Viña del Mar
- China (16):
  - Research Site, Beijing
  - Research Site, Chongqing
  - Research Site, Chuangchun
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hong Kong
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shijiazhuang
  - Research Site, Siping
  - Research Site, Suzhou
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yinchuan
- Colombia (6):
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Bogotá D.C.
  - Research Site, Cali
  - Research Site, Manizales
  - Research Site, Medellín
- Czechia (5):
  - Research Site, Olomouc-Lazce
  - Research Site, Prague
  - Research Site, Praha 10, Prague
  - Research Site, Svitavy
  - Research Site, Znojmo
- Germany (30):
  - Research Site, Aachen
  - Research Site, Aschaffenburg
  - Research Site, Bad Nauheim
  - Research Site, Bad Oeynhausen
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Burg
  - Research Site, Burghausen
  - Research Site, Chemnitz
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Eschweiler
  - Research Site, Essen
  - Research Site, Giessen
  - Research Site, Herne
  - Research Site, Hohenmölsen
  - Research Site, Kassel
  - Research Site, Kiel-Kronshagen
  - Research Site, Köthen
  - Research Site, Lichtenfels
  - Research Site, Mainz
  - Research Site, Mayen
  - Research Site, München
  - Research Site, Münster
  - Research Site, Obermichelbach
  - Research Site, Osnabrück
  - Research Site, Riesa
  - Research Site, Rotenburg (Wümme)
  - Research Site, Stuttgart
  - Research Site, Würzburg
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- Hungary (24):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Csongrád
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Győr
  - Research Site, Hódmezővásárhely
  - Research Site, Jászberény
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Komárom
  - Research Site, Mosonmagyaróvár
  - Research Site, Nagykanizsa
  - Research Site, Nyíregyháza
  - Research Site, Pápa
  - Research Site, Pécs
  - Research Site, Sátoraljaújhely
  - Research Site, Szekszárd
  - Research Site, Szentes
  - Research Site, Székesfehérvár
  - Research Site, Szigetvár
  - Research Site, Szikszó
  - Research Site, Veszprém
  - Research Site, Zalaegerszeg
- Israel (11):
  - Research Site, Giv‘atayim
  - Research Site, Hadera
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Nazareth
  - Research Site, Petah Tikva
  - Research Site, Safed
  - Research Site, Tel Aviv
- Italy (8):
  - Research Site, Florence
  - Research Site, Foggia
  - Research Site, Milan
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Sesto San Giovanni
  - Research Site, Terni
  - Research Site, Udine
- Latvia (7):
  - Research Site, Daugavpils
  - Research Site, Jelgava
  - Research Site, Kuldīga
  - Research Site, Ogre
  - Research Site, Riga
  - Research Site, Talsi
  - Research Site, Tukums
- Lithuania (7):
  - Research Site, Kaunas
  - Research Site, Kėdainiai
  - Research Site, Klaipėda
  - Research Site, Panevezys
  - Research Site, Ukmerge
  - Research Site, Utena
  - Research Site, Vilnius
- Malaysia (7):
  - Research Site, Alor Star
  - Research Site, Batu Caves
  - Research Site, Kota Samarahan
  - Research Site, Kuala Lumpur
  - Research Site, Kuching
  - Research Site, Sungai Buloh
  - Research Site, Taiping
- Mexico (9):
  - Research Site, Aguascalientes
  - Research Site, Cuautla
  - Research Site, Durango
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Puebla City
  - Research Site, Querétaro
  - Research Site, San Luis Potosí City
- Netherlands (10):
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, Eindhoven
  - Research Site, Groningen
  - Research Site, Hardenberg
  - Research Site, Hoogeveen
  - Research Site, Meppel
  - Research Site, Rotterdam
  - Research Site, Sneek
  - Research Site, Utrecht
- New Zealand (8):
  - Research Site, Christchurch
  - Research Site, Hamilton
  - Research Site, Nelson
  - Research Site, Newtown
  - Research Site, Palmerston North
  - Research Site, Takapuna
  - Research Site, Tauranga
  - Research Site, Wellington
- Philippines (8):
  - Research Site, Cebu
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Marikina City
  - Research Site, Pasig
  - Research Site, Quezon
  - Research Site, Quezon City
  - Research Site, San Juan City
- Poland (14):
  - Research Site, Elblag
  - Research Site, Gdynia
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Grudziądz
  - Research Site, Katowice
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Ostrołęka
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Słupsk
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Łęczna
- Romania (11):
  - Research Site, Bacau
  - Research Site, Bucharest
  - Research Site, Buzău
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Ploieşti
  - Research Site, Satu Mare
  - Research Site, Timișoara
  - Research Site, Zalău
- Russia (12):
  - Research Site, Kemerovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Saint Peterburg
  - Research Site, Saint Petersburg
  - Research Site, St.Рetersburg
  - Research Site, Thymen
  - Research Site, Tomsk
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg
- Slovakia (8):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Prešov
  - Research Site, Rožňava
  - Research Site, Trebišov
  - Research Site, Žilina
- South Africa (17):
  - Research Site, Boksburg
  - Research Site, Brits
  - Research Site, Cape Town
  - Research Site, Centurion
  - Research Site, Durban
  - Research Site, eMkhomazi
  - Research Site, Johannesburg
  - Research Site, Kempton Park
  - Research Site, Lenasia
  - Research Site, Paarl
  - Research Site, Parktown
  - Research Site, Phoenix
  - Research Site, Port Elizabeth
  - Research Site, Potchefstroom
  - Research Site, Pretoria
  - Research Site, Somerset West
  - Research Site, Soweto
- South Korea (9):
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Gwangjin-gu
  - Research Site, Gyeonggi-do
  - Research Site, Incheon
  - Research Site, Seongnam
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Ulsan
- Spain (15):
  - Research Site, A Coruña
  - Research Site, Alcalá de Henares
  - Research Site, Ávila
  - Research Site, Ferrol
  - Research Site, Girona
  - Research Site, Granada
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Manacor
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Palma deMallorca
  - Research Site, Salamanca
  - Research Site, Seville
  - Research Site, Tarragona
- Taiwan (8):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Kaohsiung Hsien
  - Research Site, Kweishan Shiang
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan County
  - Research Site, Taipei
- Research Site, Bangkok, Thailand
- Ukraine (17):
  - Research Site, Chernivtsi
  - Research Site, Dnipro
  - Research Site, Dnipropetrovsk
  - Research Site, Donetck
  - Research Site, Donetsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kiev
  - Research Site, Kyiv
  - Research Site, Odesa
  - Research Site, Sumy
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zaporizhia
  - Research Site, Zaporizhzhya
  - Research Site, Zhytomyr
- United Kingdom (28):
  - Research Site, Aberdeen
  - Research Site, Addlestone
  - Research Site, Birmingham
  - Research Site, Blackpool
  - Research Site, Bradford
  - Research Site, Bristol
  - Research Site, Cambridge
  - Research Site, Chippenham
  - Research Site, Coventry
  - Research Site, Dundee
  - Research Site, Edinburgh
  - Research Site, Glasgow
  - Research Site, Hull
  - Research Site, Inverness
  - Research Site, Irvine
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, Manchester
  - Research Site, Northampton
  - Research Site, Ormskirk
  - Research Site, Peterborough
  - Research Site, Plymouth
  - Research Site, Redhill
  - Research Site, Sheffield
  - Research Site, Suffolk
  - Research Site, Swansea
  - Research Site, Trowbridge
  - Research Site, West Sussex

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Koychev I, Reid G, Nguyen M, Mentz RJ, Joyce D, Shah SH, Holman RR. Inflammatory proteins associated with Alzheimer's disease reduced by a GLP1 receptor agonist: a post hoc analysis of the EXSCEL randomized placebo controlled trial. Alzheimers Res Ther. 2024 Oct 2;16(1):212. doi: 10.1186/s13195-024-01573-x. PMID 39358806
- [Derived] Gao N, Dakin HA, Holman RR, Lim LL, Leal J, Clarke P. Estimating Risk Factor Time Paths Among People with Type 2 Diabetes and QALY Gains from Risk Factor Management. Pharmacoeconomics. 2024 Sep;42(9):1017-1028. doi: 10.1007/s40273-024-01398-4. Epub 2024 Jun 26. PMID 38922488
- [Derived] Davis TME, Giczewska A, Lokhnygina Y, Mentz RJ, Sattar N, Holman RR; EXSCEL Study Group. Effect of race on cardiometabolic responses to once-weekly exenatide: insights from the Exenatide Study of Cardiovascular Event Lowering (EXSCEL). Cardiovasc Diabetol. 2022 Jun 27;21(1):116. doi: 10.1186/s12933-022-01555-z. PMID 35761271
- [Derived] Becker F, Dakin HA, Reed SD, Li Y, Leal J, Gustavson SM, Wittbrodt E, Hernandez AF, Gray AM, Holman RR. Lifetime cost-effectiveness simulation of once-weekly exenatide in type 2 diabetes: A cost-utility analysis based on the EXSCEL trial. Diabetes Res Clin Pract. 2022 Jan;183:109152. doi: 10.1016/j.diabres.2021.109152. Epub 2021 Nov 20. PMID 34813910
- [Derived] Bethel MA, Stevens SR, Buse JB, Choi J, Gustavson SM, Iqbal N, Lokhnygina Y, Mentz RJ, Patel RA, Ohman P, Schernthaner G, Lecube A, Hernandez AF, Holman RR. Exploring the Possible Impact of Unbalanced Open-Label Drop-In of Glucose-Lowering Medications on EXSCEL Outcomes. Circulation. 2020 Apr 28;141(17):1360-1370. doi: 10.1161/CIRCULATIONAHA.119.043353. Epub 2020 Feb 26. PMID 32098501
- [Derived] Standl E, Stevens SR, Lokhnygina Y, Bethel MA, Buse JB, Gustavson SM, Maggioni AP, Mentz RJ, Hernandez AF, Holman RR; EXSCEL Study Group. Confirming the Bidirectional Nature of the Association Between Severe Hypoglycemic and Cardiovascular Events in Type 2 Diabetes: Insights From EXSCEL. Diabetes Care. 2020 Mar;43(3):643-652. doi: 10.2337/dc19-1079. Epub 2019 Dec 27. PMID 31882409
- [Derived] Reed SD, Li Y, Dakin HA, Becker F, Leal J, Gustavson SM, Kartman B, Wittbrodt E, Mentz RJ, Pagidipati NJ, Bethel MA, Gray AM, Holman RR, Hernandez AF; EXSCEL Study Group. Within-Trial Evaluation of Medical Resources, Costs, and Quality of Life Among Patients With Type 2 Diabetes Participating in the Exenatide Study of Cardiovascular Event Lowering (EXSCEL). Diabetes Care. 2020 Feb;43(2):374-381. doi: 10.2337/dc19-0950. Epub 2019 Dec 5. PMID 31806653
- [Derived] Badjatiya A, Merrill P, Buse JB, Goodman SG, Katona B, Iqbal N, Pagidipati NJ, Sattar N, Holman RR, Hernandez AF, Mentz RJ, Patel MR, Jones WS. Clinical Outcomes in Patients With Type 2 Diabetes Mellitus and Peripheral Artery Disease: Results From the EXSCEL Trial. Circ Cardiovasc Interv. 2019 Dec;12(12):e008018. doi: 10.1161/CIRCINTERVENTIONS.119.008018. Epub 2019 Nov 22. PMID 31752517
- [Derived] Clegg LE, Penland RC, Bachina S, Boulton DW, Thuresson M, Heerspink HJL, Gustavson S, Sjostrom CD, Ruggles JA, Hernandez AF, Buse JB, Mentz RJ, Holman RR. Effects of exenatide and open-label SGLT2 inhibitor treatment, given in parallel or sequentially, on mortality and cardiovascular and renal outcomes in type 2 diabetes: insights from the EXSCEL trial. Cardiovasc Diabetol. 2019 Oct 22;18(1):138. doi: 10.1186/s12933-019-0942-x. PMID 31640705
- [Derived] Fudim M, White J, Pagidipati NJ, Lokhnygina Y, Wainstein J, Murin J, Iqbal N, Ohman P, Lopes RD, Reicher B, Holman RR, Hernandez AF, Mentz RJ. Effect of Once-Weekly Exenatide in Patients With Type 2 Diabetes Mellitus With and Without Heart Failure and Heart Failure-Related Outcomes: Insights From the EXSCEL Trial. Circulation. 2019 Nov 12;140(20):1613-1622. doi: 10.1161/CIRCULATIONAHA.119.041659. Epub 2019 Sep 23. PMID 31542942
- [Derived] Bethel MA, Patel RA, Thompson VP, Merrill P, Reed SD, Li Y, Ahmadi S, Katona BG, Gustavson SM, Ohman P, Iqbal N, Gagel RF, Hernandez AF, Buse JB, Holman RR; EXSCEL Study Group. Changes in Serum Calcitonin Concentrations, Incidence of Medullary Thyroid Carcinoma, and Impact of Routine Calcitonin Concentration Monitoring in the EXenatide Study of Cardiovascular Event Lowering (EXSCEL). Diabetes Care. 2019 Jun;42(6):1075-1080. doi: 10.2337/dc18-2028. Epub 2019 Apr 22. PMID 31010875
- [Derived] Mentz RJ, Bethel MA, Merrill P, Lokhnygina Y, Buse JB, Chan JC, Felicio JS, Goodman SG, Choi J, Gustavson SM, Iqbal N, Lopes RD, Maggioni AP, Ohman P, Pagidipati NJ, Poulter NR, Ramachandran A, Reicher B, Holman RR, Hernandez AF; EXSCEL Study Group. Effect of Once-Weekly Exenatide on Clinical Outcomes According to Baseline Risk in Patients With Type 2 Diabetes Mellitus: Insights From the EXSCEL Trial. J Am Heart Assoc. 2018 Oct 2;7(19):e009304. doi: 10.1161/JAHA.118.009304. PMID 30371301
- [Derived] Wittbrodt ET, Eudicone JM, Bell KF, Enhoffer DM, Latham K, Green JB. Generalizability of glucagon-like peptide-1 receptor agonist cardiovascular outcome trials enrollment criteria to the US type 2 diabetes population. Am J Manag Care. 2018 Apr;24(8 Suppl):S146-S155. PMID 29693361
- [Derived] Holman RR, Bethel MA, Mentz RJ, Thompson VP, Lokhnygina Y, Buse JB, Chan JC, Choi J, Gustavson SM, Iqbal N, Maggioni AP, Marso SP, Ohman P, Pagidipati NJ, Poulter N, Ramachandran A, Zinman B, Hernandez AF; EXSCEL Study Group. Effects of Once-Weekly Exenatide on Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2017 Sep 28;377(13):1228-1239. doi: 10.1056/NEJMoa1612917. Epub 2017 Sep 14. PMID 28910237
- [Derived] Mentz RJ, Bethel MA, Gustavson S, Thompson VP, Pagidipati NJ, Buse JB, Chan JC, Iqbal N, Maggioni AP, Marso SP, Ohman P, Poulter N, Ramachandran A, Zinman B, Hernandez AF, Holman RR. Baseline characteristics of patients enrolled in the Exenatide Study of Cardiovascular Event Lowering (EXSCEL). Am Heart J. 2017 May;187:1-9. doi: 10.1016/j.ahj.2017.02.005. Epub 2017 Feb 12. PMID 28454792
- [Derived] Holman RR, Bethel MA, George J, Sourij H, Doran Z, Keenan J, Khurmi NS, Mentz RJ, Oulhaj A, Buse JB, Chan JC, Iqbal N, Kundu S, Maggioni AP, Marso SP, Ohman P, Pencina MJ, Poulter N, Porter LE, Ramachandran A, Zinman B, Hernandez AF. Rationale and design of the EXenatide Study of Cardiovascular Event Lowering (EXSCEL) trial. Am Heart J. 2016 Apr;174:103-10. doi: 10.1016/j.ahj.2015.12.009. Epub 2015 Dec 21. PMID 26995376
- [Derived] Gaebler JA, Soto-Campos G, Alperin P, Cohen M, Blickensderfer A, Wintle M, Maggs D, Hoogwerf B, Han J, Pencek R, Peskin B. Health and economic outcomes for exenatide once weekly, insulin, and pioglitazone therapies in the treatment of type 2 diabetes: a simulation analysis. Vasc Health Risk Manag. 2012;8:255-64. doi: 10.2147/VHRM.S28744. Epub 2012 Apr 23. PMID 22566747
- See also: d5551c00003_bcb109_csp_amendment_6_updated_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3675&filename=d5551c00003_bcb109_csp_amendment_6_updated_Redacted.pdf
- See also: d5551c00003 SAP Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3675&filename=d5551c00003_SAP_Redacted.pdf
- See also: d5551c00003 CSP Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3675&filename=d5551c00003_CSP_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo subcutaneous injections
- Exenatide Once Weekly: Exenatide 2mg once weekly subcutaneous injections
Period: Overall Study
Arm/Group | Placebo | Exenatide Once Weekly
Started | 7396 | 7356
Completed | 7093 | 7094
Not Completed | 303 | 262

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Exenatide Once Weekly | Total
Number analyzed (Participants) | 7396 | 7356 | 14752
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at enrollment
  Years | 61.9 (9.4) | 61.8 (9.4) | 61.9 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2809 | 2794 | 5603
  Male | 4587 | 4562 | 9149
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 5621 | 5554 | 11175
  BLACK OR AFRICAN AMERICAN | 436 | 442 | 878
  ASIAN | 727 | 725 | 1452
  INDIAN (AMERICAN ) OR ALASKA NATIVE | 35 | 38 | 73
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 17 | 18 | 35
  HISPANIC | 557 | 577 | 1134
  MISSING | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Global: ASIA PACIFIC | 760 | 769 | 1529
  Global: EUROPE | 3399 | 3389 | 6788
  Global: LATIN AMERICA | 1363 | 1364 | 2727
  Global: NORTH AMERICA | 1874 | 1834 | 3708
Prior CV Event [Count of Participants; unit: Participants] — Patient had prior cardiovascular event or not at randomization
  Participants
    Yes | 5388 | 5394 | 10782
    No | 2008 | 1962 | 3970

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Outcome MACE Events
Description: The primary efficacy outcome variable is defined as the composite endpoint of cardiovascular death, nonfatal MI, or nonfatal stroke. The number of participants who had an event is reported in the results.
  The primary efficacy endpoint is the same as the primary safety endpoint, and the statistical analysis tests the superiority of exenatide against the placebo.
Time Frame: Time to first event. Information collected during study period (anticipated to be up to 7.5 years).
Population: ITT population: all patients consented and randomized in the study without a major GCP violation. ITT population is analyzed as randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Exenatide Once Weekly
Number analyzed (Participants) | 7396 | 7356
Participants
  Number of patients who had a MACE event | 905 | 839
Statistical Analysis 1: Comparison: Placebo vs Exenatide Once Weekly; Test type: Superiority — Superiority test of EQW over Placebo H0: HR ≥ 1 vs. H1: HR < 1; p = 0.061, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.832 to 1.004]

2. Primary Outcome: Primary Safety Outcome MACE Events
Description: The primary safety outcome variable is defined as the composite endpoint of cardiovascular death, nonfatal MI, or nonfatal stroke. The number of participants who had an event is reported in the results.
  The primary safety endpoint is the same as the primary efficacy endpoints, and the statistical analysis tests the non-inferiority of exenatide against placebo.
Time Frame: Time to first event. Information collected during study period (anticipated to be up to 7.5 years).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Exenatide Once Weekly
Number analyzed (Participants) | 7396 | 7356
Participants
  Number of patients who had a MACE event | 905 | 839
Statistical Analysis 1: Comparison: Placebo vs Exenatide Once Weekly; This analysis uses the same endpoint and cox regression method as the primary efficacy analysis. However, the statistical hypothesis is a non-inferiority test with a margin of HR=1.3; Test type: Non-Inferiority — Non-inferiority test of EQW over Placebo H0: HR ≥ 1.3 vs. H1: HR < 1.3; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.832 to 1.004]

3. Secondary Outcome: Secondary Efficacy Outcome All-Cause Mortality
Description: The secondary efficacy outcome variable is defined as the all-cause mortality (deaths). The number of participants who had an event is reported in the results.
Time Frame: Time to first event. Information collected during study period (anticipated to be up to 7.5 years).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Exenatide Once Weekly
Number analyzed (Participants) | 7396 | 7356
Participants
  Number of patients who died | 584 | 507
Statistical Analysis 1: Comparison: Placebo vs Exenatide Once Weekly; Test type: Superiority — Superiority test of EQW over Placebo H0: HR ≥ 1 vs. H1: HR < 1; p = 0.016, Regression, Cox; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.77 to 0.97]

4. Secondary Outcome: Secondary Efficacy Outcome CV Death
Description: Component of the primary efficacy outcome: cardiovascular death. The number of participants who had an event is reported in the results.
Time Frame: Time to first event. Information collected during study period (anticipated to be up to 7.5 years).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Exenatide Once Weekly
Number analyzed (Participants) | 7396 | 7356
Participants
  Number of patients who had CV death | 383 | 340
Statistical Analysis 1: Comparison: Placebo vs Exenatide Once Weekly; Test type: Superiority — Superiority test of EQW over Placebo H0: HR ≥ 1 vs. H1: HR < 1; p = 0.096, Regression, Cox; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.76 to 1.02]

5. Secondary Outcome: Secondary Efficacy Outcome MI
Description: Component of primary efficacy outcome: fatal or non-fatal MI. The number of participants who had an event is reported in the results.
Time Frame: Time to first event. Information collected during study period (anticipated to be up to 7.5 years).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Exenatide Once Weekly
Number analyzed (Participants) | 7396 | 7356
Participants
  Number of patients who died | 493 | 483
Statistical Analysis 1: Comparison: Placebo vs Exenatide Once Weekly; Test type: Superiority — Superiority test of EQW over Placebo H0: HR ≥ 1 vs. H1: HR < 1; p = 0.622, Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.85 to 1.10]

6. Secondary Outcome: Secondary Efficacy Outcome Stroke
Description: Component of primary efficacy outcome: fatal or non-fatal stroke. The number of participants who had an event is reported in the results.
Time Frame: Time to first event. Information collected during study period (anticipated to be up to 7.5 years).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Exenatide Once Weekly
Number analyzed (Participants) | 7396 | 7356
Participants
  Number of patients who had stroke | 218 | 187
Statistical Analysis 1: Comparison: Placebo vs Exenatide Once Weekly; Test type: Superiority — Superiority test of EQW over Placebo H0: HR ≥ 1 vs. H1: HR < 1; p = 0.095, Regression, Cox; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.70 to 1.03]

7. Secondary Outcome: Secondary Efficacy Outcome Hospitalization for ACS
Description: The secondary efficacy outcome variable is defined as hospitalization for acute coronary syndrome. The number of participants who had an event is reported in the results.
Time Frame: Time to first event. Information collected during study period (anticipated to be up to 7.5 years).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Exenatide Once Weekly
Number analyzed (Participants) | 7396 | 7356
Participants
  Num of pts with hospitalization due to ACS | 570 | 602
Statistical Analysis 1: Comparison: Placebo vs Exenatide Once Weekly; Test type: Superiority — Superiority test of EQW over Placebo H0: HR ≥ 1 vs. H1: HR < 1; p = 0.402, Regression, Cox; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.94 to 1.18]

8. Secondary Outcome: Secondary Efficacy Outcome Hospitalization for HF
Description: The secondary efficacy outcome variable is defined as hospitalization for heart failure. The number of participants who had an event is reported in the results.
Time Frame: Time to first event. Information collected during study period (anticipated to be up to 7.5 years).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Exenatide Once Weekly
Number analyzed (Participants) | 7396 | 7356
Participants
  Number of patients who died | 231 | 219
Statistical Analysis 1: Comparison: Placebo vs Exenatide Once Weekly; Test type: Superiority — Superiority test of EQW over Placebo H0: HR ≥ 1 vs. H1: HR < 1; p = 0.485, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.78 to 1.13]

ADVERSE EVENTS:
Time Frame: During study period up to 7.5 years
Description: Only SAEs are collected in this study. Other (not including non-serious) adverse events are not monitored/assessed.
Arm/Group | Placebo | Exenatide Once Weekly
All-Cause Mortality (participants affected / at risk) | 584/7372 | 507/7344
Serious Adverse Events (participants affected / at risk) | 1222/7372 | 1234/7344
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7372) | Exenatide Once Weekly (N=7344)
Anaemia (Blood and lymphatic system disorders) | 26 (31) | 15 (16)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow oedema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 11 (13)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mastocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 3 (3) | 0 (0)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 1 (2) | 0 (0)
Sacralisation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Thalassaemia beta (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Mixed deafness (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 6 (6) | 6 (7)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 6 (6)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Cushing's syndrome (Endocrine disorders) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 3 (4) | 7 (7)
Hyperaldosteronism (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 2 (3) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Thyroid disorder (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 2 (2)
Extraocular muscle disorder (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 1 (2) | 1 (1)
Lens dislocation (Eye disorders) | 0 (0) | 1 (1)
Macular fibrosis (Eye disorders) | 0 (0) | 1 (1)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Macular oedema (Eye disorders) | 1 (1) | 0 (0)
Open angle glaucoma (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 3 (3) | 4 (4)
Retinal haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 2 (2) | 3 (3)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (2)
Abdominal hernia (Gastrointestinal disorders) | 6 (6) | 7 (7)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2)
Abdominal strangulated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (2) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anorectal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorectal varices (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 2 (2) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 1 (2)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 2 (2) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 (3) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 2 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Enterocele (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Erosive oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4)
Gastric ulcer perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 12 (12) | 4 (4)
Gastritis erosive (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 34 (37) | 27 (30)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal melanosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 (10) | 6 (8)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 3 (3)
Ileus (Gastrointestinal disorders) | 2 (2) | 3 (3)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Inflammatory bowel disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 4 (4) | 9 (9)
Intestinal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 4 (4)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 10 (11) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 (9) | 3 (4)
Lumbar hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Mallory-weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oroantral fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 22 (24) | 37 (37)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peritoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (3) | 5 (5)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectourethral fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 8 (9) | 7 (7)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Subileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tongue haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 14 (14) | 5 (5)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 (10) | 9 (9)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 5 (5) | 4 (4)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 5 (5) | 5 (5)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1)
Drug interaction (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 2 (2)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 2 (2)
Granuloma (General disorders) | 1 (1) | 1 (1)
Haemorrhagic cyst (General disorders) | 0 (0) | 1 (1)
Hernia (General disorders) | 2 (2) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Impaired self-care (General disorders) | 0 (0) | 1 (2)
Injection site inflammation (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 3 (3)
Non-cardiac chest pain (General disorders) | 79 (90) | 87 (104)
Oedema (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1)
Polyp (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 0 (0)
Strangulated hernia (General disorders) | 0 (0) | 2 (2)
Acute hepatic failure (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biliary cyst (Hepatobiliary disorders) | 1 (1) | 0 (0)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (3) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder fistula (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 3 (3) | 4 (5)
Hepatic haematoma (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatosplenomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 3 (3)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic tonsillitis (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis e (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2) | 1 (1)
Herpes zoster oticus (Infections and infestations) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Keratouveitis (Infections and infestations) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 7 (7) | 11 (11)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Complicated fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Contrast media reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Ear injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 14 (15) | 12 (12)
Femoral neck fracture (Injury, poisoning and procedural complications) | 6 (6) | 10 (10)
Femur fracture (Injury, poisoning and procedural complications) | 13 (14) | 9 (9)
Fibula fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Forearm fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haematuria traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 6 (6) | 14 (14)
Humerus fracture (Injury, poisoning and procedural complications) | 9 (10) | 10 (10)
Ilium fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Lower limb fracture (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Meniscus injury (Injury, poisoning and procedural complications) | 7 (7) | 6 (7)
Multiple fractures (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 7 (7) | 5 (5)
Patella fracture (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Perirenal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 14 (14) | 5 (5)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Scapula fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skull fractured base (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal column injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Splenic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 9 (9) | 11 (11)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 8 (8) | 8 (8)
Toxicity to various agents (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Upper limb fracture (Injury, poisoning and procedural complications) | 3 (3) | 7 (7)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound evisceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 2 (3) | 3 (3)
Anticoagulation drug level increased (Investigations) | 1 (1) | 0 (0)
Blood calcitonin increased (Investigations) | 0 (0) | 1 (1)
Blood potassium decreased (Investigations) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1)
Hiv test positive (Investigations) | 1 (1) | 0 (0)
International normalised ratio abnormal (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 3 (3)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 10 (10)
Electrolyte imbalance (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 8 (9)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 9 (10) | 1 (1)
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Articular calcification (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (14) | 14 (15)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Chest wall haematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Crystal arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Deformity thorax (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (5)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 17 (19) | 15 (18)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint adhesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 20 (21) | 12 (13)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Monarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 10 (13)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 79 (89) | 69 (76)
Osteochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Periostitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 9 (9) | 5 (5)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 10 (10) | 4 (4)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 11 (13)
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acth-producing pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 12 (12)
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Appendix cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 (33) | 25 (42)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign small intestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 9 (9)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (6)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (14) | 16 (16)
Breast cancer male (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid body tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Clear cell endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 16 (16)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Colon cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Desmoplastic melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large b-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
Endometrial adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (4)
Epithelioid mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Extradural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (5)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal submucosal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hairy cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 2 (2)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (2)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (4)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 6 (6)
Lung carcinoma cell type unspecified stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 (12) | 12 (12)
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Malignant anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 8 (8)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Non-small cell lung cancer stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15) | 15 (15)
Pancreatic neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Paraproteinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Peripheral t-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 5 (5)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 (26) | 20 (20)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 2 (2)
Prostate cancer stage i (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 5 (5)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Respiratory papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Retinal melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Spinal meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (16) | 12 (15)
Squamous cell carcinoma of head and neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 7 (8)
Squamous cell carcinoma of the hypopharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 14 (14)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 5 (5)
Transitional cell carcinoma urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Xanthogranuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 2 (2) | 1 (1)
Amputation stump pain (Nervous system disorders) | 0 (0) | 1 (1)
Asterixis (Nervous system disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 2 (2) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Brain injury (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 4 (5) | 5 (5)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 5 (5) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 2 (2) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 1 (1) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 3 (3) | 0 (0)
Cervicogenic headache (Nervous system disorders) | 1 (1) | 1 (1)
Cognitive disorder (Nervous system disorders) | 2 (2) | 0 (0)
Coma (Nervous system disorders) | 1 (1) | 1 (1)
Coordination abnormal (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 2 (2) | 2 (2)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 3 (3)
Demyelinating polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 9 (9) | 5 (6)
Encephalopathy (Nervous system disorders) | 4 (5) | 4 (4)
Epilepsy (Nervous system disorders) | 2 (2) | 5 (5)
Facial paralysis (Nervous system disorders) | 6 (6) | 4 (4)
Facial paresis (Nervous system disorders) | 1 (1) | 1 (1)
Frontotemporal dementia (Nervous system disorders) | 0 (0) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-barre syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 2 (2)
Hepatic encephalopathy (Nervous system disorders) | 3 (5) | 4 (5)
Hydrocephalus (Nervous system disorders) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1)
Iiird nerve paralysis (Nervous system disorders) | 0 (0) | 3 (3)
Idiopathic generalised epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 3 (3)
Lumbosacral radiculopathy (Nervous system disorders) | 1 (1) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 2 (2)
Migraine (Nervous system disorders) | 2 (2) | 6 (6)
Mixed dementia (Nervous system disorders) | 1 (1) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 3 (3)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Nerve root compression (Nervous system disorders) | 1 (1) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 2 (2)
Neuralgic amyotrophy (Nervous system disorders) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 1 (1) | 0 (0)
Neurodegenerative disorder (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 2 (2)
Normal pressure hydrocephalus (Nervous system disorders) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Parkinsonism (Nervous system disorders) | 0 (0) | 2 (2)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Post stroke seizure (Nervous system disorders) | 1 (1) | 0 (0)
Radicular syndrome (Nervous system disorders) | 1 (1) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 4 (4)
Seizure (Nervous system disorders) | 10 (10) | 6 (7)
Senile dementia (Nervous system disorders) | 0 (0) | 1 (1)
Spinal claudication (Nervous system disorders) | 1 (1) | 1 (1)
Spinal cord compression (Nervous system disorders) | 2 (2) | 1 (1)
Spondylitic myelopathy (Nervous system disorders) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 3 (3) | 0 (0)
Subacute combined cord degeneration (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Subdural hygroma (Nervous system disorders) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Vith nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 2 (2) | 1 (1)
Vascular headache (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 4 (5) | 2 (2)
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Cephalo-pelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Device battery issue (Product Issues) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 3 (3)
Device failure (Product Issues) | 0 (0) | 1 (1)
Device loosening (Product Issues) | 3 (3) | 3 (3)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 1 (1)
Patient-device incompatibility (Product Issues) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 2 (3) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 14 (15) | 6 (7)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 2 (2) | 3 (3)
Mental status changes (Psychiatric disorders) | 0 (0) | 7 (7)
Personality change due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Psychogenic seizure (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (2) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 2 (2)
Suicide attempt (Psychiatric disorders) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Azotaemia (Renal and urinary disorders) | 2 (2) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder diverticulum (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 2 (2) | 0 (0)
Calculus urethral (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 5 (5) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis chronic (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 7 (7) | 6 (6)
Hydronephrosis (Renal and urinary disorders) | 4 (5) | 1 (1)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypotonic urinary bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 13 (13) | 15 (16)
Nephrosclerosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 3 (3) | 8 (8)
Renal cyst (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureteric stenosis (Renal and urinary disorders) | 3 (3) | 1 (2)
Ureterolithiasis (Renal and urinary disorders) | 5 (5) | 10 (10)
Urethral haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 3 (3)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 7 (8) | 4 (4)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 2 (2)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 11 (11) | 9 (9)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital lesion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Organic erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 3 (3) | 2 (2)
Ovarian vein thrombosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 8 (8)
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 5 (6)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 49 (81) | 48 (84)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 11 (13)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal septum perforation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (10)
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 12 (13)
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 7 (7)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 5 (7) | 5 (5)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Parapsoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Prurigo (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Umbilical haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Alcohol use (Social circumstances) | 1 (1) | 0 (0)
Arterial rupture (Vascular disorders) | 1 (1) | 0 (0)
Bleeding varicose vein (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 8 (8)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Post thrombotic syndrome (Vascular disorders) | 0 (0) | 1 (1)
Temporal arteritis (Vascular disorders) | 1 (2) | 0 (0)
Varicose vein (Vascular disorders) | 3 (3) | 2 (2)

LIMITATIONS AND CAVEATS:
Only SAE are collected in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2009-12-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT01144338/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-23): https://cdn.clinicaltrials.gov/large-docs/38/NCT01144338/SAP_001.pdf